CLINICAL TRIAL: NCT01823094
Title: CTP (Computed Tomography Perfusion) Imaging of Lung Cancer
Brief Title: CTP Imaging of Lung Cancer
Acronym: CTPLC
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Collaborators: Radiological Society of North America (Other)
Responsible Party: Sponsor
Other Study IDs: 393991
Record Dates: First submitted 2013-03-22; First posted 2013-04-04 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Non Small Cell Lung Cancer
Keywords: lung cancer; computed tomography; blood flow
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Variability of measurements: variability of CTP measurements will be determined by repeating the CTP examination, and comparing the resultant blood flow estimates
- Treatment induced effects: The magnitude of treatment induced effects will be assessed by comparing tumor blood flow estimates before and after treatment

SUMMARY:
Investigators hope to learn more about how to use computed tomography (CT) scans to measure blood flow in lung tumors and how it may change in response to treatment. This measurement technique is called computed tomography perfusion (CTP). CT scanners use X-rays to produce 3-dimensional images of the body.

Currently, doctors determine the response to treatment by measuring the size of the tumor. Investigators are trying to find out if measuring the blood flow in the tumor is equal to or better than measuring the size of the tumor.

DETAILED DESCRIPTION:
This is an experimental study of CT perfusion (CTP) imaging in subjects with non-small cell lung cancer. The objectives of this study are to demonstrate the feasibility of CT blood flow measurements in lung cancer, to develop a foundation for the use of CT blood flow measurements in lung cancer to assess the response to treatment, and to develop an optimized CTP imaging protocol for evaluating blood flow in solid body tumors. In this study, tumor blood flow will be evaluated at baseline and follow-up routine CT examinations of patients with non-small cell lung cancer, and the response of tumor blood flow will be recorded as a secondary endpoint. This research study will entail two study visits - one required and one optional - which will coincide with regularly scheduled standard of care CT scans.

ELIGIBILITY:
Inclusion Criteria:

adult patients with non small cell lung cancer who receive, or are considered for, systemic therapy

Exclusion Criteria:

renal failure pregnancy known contrast allergy

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with non small cell lung cancer who are planned to receive systemic therapy
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2013-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Yield of conducting CTP studies | 2 years
  Yield is determined as the percentage of assessable CTP studies, relative to all performed studies

SECONDARY OUTCOMES:
Variability of CTP measurements | 2 years
  Variability will be determined from two consecutively acquired CTP examinations, and repeated analyses of the same studies
Magnitude of treatment induced changes in tumor blood flow | 2 years
  The magnitude of treatment induced changes in blood flow will be determined from comparisons of bloodflow before and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Friedrich Knollmann, MD, PhD, Principal Investigator — Univeristy of California, Davis
Locations (1):
- University of California, Davis Medical Center, Sacramento, California, United States